CLINICAL TRIAL: NCT01784770
Title: Zithromac Iv Special Investigation For Legionella Infection.
Brief Title: Special Investigation Of Azithromycin IV For Legionnaires' Disease (Regulatory Post Marketing Commitment Plan)
Acronym: RESCUE-L
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0661208
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-07

CONDITIONS: Legionnaires' Disease; Legionella Pneumophila Infections
Keywords: Legionnaires' disease; Legionella pneumophila; Zithromax; Zithromac; Japanese; Regulatory Post Marketing Commitment Plan
MeSH Terms: conditions — Legionnaires' Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Azithromycin IV: Subjects who are treated with Azithromycin IV for Legionnaires' disease
  Interventions: Drug: Azithromycin IV

INTERVENTIONS:
Drug: Azithromycin IV — The recommended dose of ZITHROMAC (azithromycin for injection) for the treatment of adult patients with community-acquired pneumonia due to the indicated organisms is: 500 mg as a single daily dose by the intravenous route for at least two days. Intravenous therapy should be followed by azithromycin by the oral route at a single, daily dose of 500 mg, administered as two 250-mg tablets to complete a 7- to 10-day course of therapy.
  The recommended dose of ZITHROMAC (azithromycin for injection) for the treatment of adult patients with pelvic inflammatory disease due to the indicated organisms is: 500 mg as a single daily dose by the intravenous route for one or two days. Intravenous therapy should be followed by azithromycin by the oral route at a single, daily dose of 250 mg to complete a 7-day course of therapy.
  Other Names: Zithromac IV

SUMMARY:
To collect retrospectively the efficacy and safety information of azithromycin IV on patients with Legionnaires' disease related to their appropriate use in daily practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are prescribed Azithromycin (Zithromac) IV for Legionnaires' disease.

Exclusion Criteria:

* Patients who have been prescribed Zithromac or Zithromac SR.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A0661208 prescribes the Zithromac IV.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-03-27 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661208&StudyName=Special%20Investigation%20Of%20Azithromycin%20IV%20For%20Legionnaires%27%20Disease%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Zithromac Intravenous Use (Azithromycin Hydrate): Participants who received Zithromac Intravenous use (and Zithromac Tablets) as indicated in the approved local product document were observed for a period of 29 days. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Zithromac Intravenous Use (Azithromycin Hydrate)
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 21 participants completed this study. There is no protocol violation.
Arm/Group | Zithromac Intravenous Use (Azithromycin Hydrate)
Number analyzed (Participants) | 21
Age, Customized [Number; unit: Participants]
  <15 years | 0
  ≥15 and <65 years | 14
  ≥65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Zithromac Intravenous use (and Zithromac Tablets) in a participant who received Zithromac Intravenous use. A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to Zithromac Intravenous use (and Zithromac Tablets) was assessed by the physician.
Time Frame: 29 days
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and received Zithromac Intravenous use at least once.
Measure: Number; unit: Participants
Arm/Group | Zithromac Intravenous Use (Azithromycin Hydrate)
Number analyzed (Participants) | 21
Participants
  Treatment-Related Adverse Event | 2
  Treatment-Related Serious Adverse Event | 0

2. Secondary Outcome: Clinical Effectiveness Rate in Participants
Description: Clinical effectiveness rate in participants, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of asssable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Clinical effectiveness of Zithromac Intravenous use (and Zithromac Tablets) was determined by the physician based on clinical symptoms and laboratory findings, and assessed according to the following categories: (1) effective, (2) ineffective, or (3) unassessable.
Time Frame: 29 days
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (overall evaluation by the physician based upon change in clinical symptoms and laboratory findings) at least once. Participants evaluated as "unassessable" were excluded from the calculation.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Zithromac Intravenous Use (Azithromycin Hydrate)
Number analyzed (Participants) | 21
Percentage of Participants | 95.2 [76.18 to 99.88]

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Zithromac Intravenous Use (Azithromycin Hydrate)
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zithromac Intravenous Use (Azithromycin Hydrate) (N=21)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zithromac Intravenous Use (Azithromycin Hydrate) (N=21)
Bradycardia (Cardiac disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1
Crystalluria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.